CLINICAL TRIAL: NCT01502449
Title: Randomized Trial of Telephonic Psychotherapy and Case Management for Combat-Related Posttraumatic Stress Disorder
Brief Title: Delivery of Self Training and Education for Stressful Situations-Telephone Version
Acronym: DESTRESS-T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Engel, Dir., Deployment Health Clinical Center; Associate Professor, psychiatry, USUHS, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D10-I-AR-J5-786
Record Dates: First submitted 2011-12-12; First posted 2011-12-30 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: PTSD
Keywords: telemedicine, telephonic, PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DESTRESS-T (Experimental): Usual primary care PTSD treatment, plus a telephone care management program over 8 weeks that includes: four outreach calls, feedback to the treating primary care provider, and care coordination
  Interventions: Behavioral: DESTRESS-T
- Optimized Usual Care (OUC) (Active Comparator): Optimized Usual Care is usual primary care PTSD treatment, plus a telephone care management program that includes: four outreach calls, feedback to the treating primary care provider (PCP), and care coordination.
  Interventions: Other: Optimized Usual Care (OUC)

INTERVENTIONS:
Behavioral: DESTRESS-T — Usual primary care PTSD treatment, plus a telephone care management program that includes: four outreach calls, feedback to the treating primary care provider, and care coordination
  Other Names: Delivery of Self-Training for Stressful Situations, Telephonic version
  Arms: DESTRESS-T
Other: Optimized Usual Care (OUC) — Optimized Usual Care is usual primary care PTSD treatment, plus a telephone care management program that includes: four outreach calls, feedback to the treating primary care provider (PCP), and care coordination.
  Arms: Optimized Usual Care (OUC)

SUMMARY:
This study will evaluate a telephone-delivered cognitive-behavioral psychotherapy intervention designed for primary care treatment of combat-exposed service members with PTSD. The investigators will assess Posttraumatic Stress Disorder (PTSD) symptoms, mental health-related and occupational functioning, and symptoms of depression, anxiety, and somatization.

DETAILED DESCRIPTION:
This is a randomized controlled trial that will compare DESTRESS-T to Optimized Usual Care (OUC). Optimized Usual Care is usual primary care PTSD treatment, plus a telephone care management program that includes: four outreach calls, feedback to the treating primary care provider (PCP), and care coordination.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* DSM-IV diagnosis of PTSD (derived from the CAPS) due to combat in OIF/OEF deployment
* Active duty personnel

Exclusion Criteria:

* Active suicidal or violent ideation within the past two months as assessed by the MINI and a supplementary form developed by the project team (see Appendices)
* Current participation in any active psychotherapy (e.g., psychoanalysis, CBT) for mood, anxiety or substance use disorders (as determined via service member self report and/or check of medical record)
* Recurrent PTSD treatment failure in psychotherapy, as determined via consensus of study team members (Dr. Charles Engel, Dr. Brett Litz, and Dr. Kristie Gore)
* Current alcohol dependence, as assessed by MINI
* Acute psychosis, psychotic episode, or psychotic disorder diagnosis within the past year, as assessed by the MINI
* Currently on an antipsychotic or mood-stabilizing agent for bipolar disorder or any disorder with psychotic features, as determined by medical record and/or self report
* Unstable administration schedule or dosing of any antidepressant, anxiolytic, or sedative-hypnotic (i.e., will exclude for any related medication changes in the month prior to randomization), as determined by medical record or service member self report
* Acute or unstable physical illness based on the judgment of the patient's primary care clinician and the study team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist - Civilian Version (PCL) | Baseline, 12 weeks, 18 weeks, and 24 weeks
  Symptoms of PTSD will be assessed using the PTSD Checklist-Civilian Version. The PCL is a self-report measure developed for measuring PTSD symptom severity and for estimating PTSD caseness when administration of a structured clinical interview is not feasible. Respondents rate PCL items on a 5-point scale ("not at all" through "extremely") to indicate the degree to which they have been bothered by each of 17 PTSD symptoms during the past month. Possible PCL scores range from 17 to 85.

SECONDARY OUTCOMES:
Medical Outcomes Survey Short-Form-12 (SF-12) | Baseline, 12 weeks, 18 weeks, and 24 weeks
  The SF-12 is a commonly used measure of mental and physical functional status. The 12 items in the SF-12 are a subset of those in the SF-36. The SF-12 contains one or two items from each of the eight health scales: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, and role limitations due to emotional problems and mental health (psychological distress and psychological well being). The SF-12 will allow us to characterize the functional status of our sample.
World Health Organization Health & Work Performance Questionnaire (HPQ) | Baseline, 12 weeks, 18 weeks, and 24 weeks
  We will use the 21-item 7-day clinical trial version of the World Health Organization Health & Work Performance Questionnaire (HPQ) to measure the impact of DESTRESS-PC on occupational functioning. The HPQ is a self-report questionnaire that obtains information about three types of workplace consequences: absenteeism (missed work days due to illness), presenteeism (low performance at work), and critical incidents.
Patient Health Questionnaire (PHQ) | Baseline, 12 weeks, 18 weeks, and 24 weeks
  The PHQ is a self-report assessment of common mental disorders developed specifically for primary care. PHQ allows brief provisional primary care diagnoses of a several disorders including major depression, panic disorder, other anxiety disorder, and multisomatoform disorder. We will use the PHQ for brief assessments of depression, anxiety (panic and generalized anxiety), and somatic symptom severity, assessments with excellent correspondence to DSM-IV diagnostic criteria.
Generalized Anxiety Symptom Severity (GAD-7) | Baseline
  Generalized anxiety symptoms will be assessed using the GAD-7, a brief measure designed for use in general health settings.
Sheehan Disability Scale (SDS) | baseline, 12 week, 18 week and 24 week
  The SDS is a three-item self-reporting tool measuring the impairment of a disability on work, social life and family life/home responsibilities. SDS is scored on a 10-point scale with 0 being "not at all disrupted" and being 10 "extremely disrupted" with any item scoring above 5 indicating a significant functional impairment in that domain. It has been used as an outcome measure in studies of PTSD due to its construct criterion related validity.
Alcohol Use Disorders Identification Test-Civilian version (AUDIT-C) | baseline, 12 week, 18 week, and 24 week
  Audit-C is a brief screen that has been found to effectively discriminate between patients with a history of drinking problems and those without such a history, including hazardous drinking. Its brevity ensures that clinicians will remember it, and administration time is minimal. A positive total score is an indication for further screening and assessment
Numeric Rating Scale for Pain (NRS). | baseline, 12 week, 18 week, and 24 week
  The NRS directs participants to rate pain intensity using three, 11-point, 0 ("no pain") to 10 ("pain as bad as you can imagine") numeric rating scales. Instructions ask participants to "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours", pain "at its worst", and "pain at its least". The NRS will be used in this study to evaluate the effect of acupuncture on comorbid symptoms of pain.

CONTACTS AND LOCATIONS:
Overall Officials: COL Charles C. Engel, MD, MPH, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Fort Benning - Martin Army Community Hospital, Columbus, Georgia, United States